CLINICAL TRIAL: NCT03126331
Title: A Single-arm Phase II Trial of Intermittent Nivolumab in Patients With Metastatic Renal Cell Carcinoma Who Have Received Prior Anti-Angiogenic Therapy
Brief Title: Intermittent Therapy in Metastatic Renal Cell Carcinoma Patients Treated With Ipilimumab and Nivolumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5816
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Kidney Cancer; Metastatic; Nivolumab
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasm Metastasis | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I: Intermittent Nivolumab (Experimental): Nivolumab monotherapy. Participants who have initial 10% or greater tumor burden reduction will discontinue nivolumab until they experience a pre-specified disease progression at which time nivolumab will be restarted
  Interventions: Drug: Nivolumab
- Cohort II: combination ipilimumab/nivolumab (Experimental): Combination of ipilimumab/nivolumab for previously untreated intermediate and poor risk mRCC
  Includes participants treated front-line ipilimumab/nivolumab. Participants with treatment-naïve mRCC who receive up to four doses of induction ipilimumab/nivolumab and 24 weeks (+/- 8 weeks; minimum 3 infusions) of maintenance nivolumab and achieve stable disease (SD), complete response (CR), or partial response (PR) will be eligible for inclusion. Participants who achieve SD will continue with nivolumab maintenance per standard of care while those who achieve a PR or CR will enter an observation period off therapy. Upon disease progression, participants will be re-challenged with combination ipilimumab/nivolumab.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab monotherapy will be administered dosed at 480mg IV over 30 minutes for all patients every 4 weeks, regardless of weight (when given in combination with ipilimumab, the dose of nivolumab is 3mg/kg every 3 weeks).
  Tumor assessed after 12 weeks If tumor decreases by 10% or more, then hold drug for 12 week and test tumor again. Continue treatment if tumor is not decreased by 10% or more.
  Other Names: Opdivo®
Drug: Ipilimumab — Ipilimumab is dosed at 1mg/kg over 30 minutes every 3 weeks
  Arms: Cohort II: combination ipilimumab/nivolumab

SUMMARY:
This study is being done with patients with advanced kidney cancer (also called renal cell carcinoma or RCC). This is a research study involving the use of the drug Nivolumab (also known as Opdivo®). Nivolumab is an anti-PD-1 antibody. It works by attaching to and blocking a molecule called PD-1. PD-1 is a protein that is present on different types of cells in the immune system and controls parts of the immune system by shutting it down. Antibodies that block PD-1 can potentially prevent PD-1 from shutting down the immune system, thus allowing it to recognize and help destroy cancer cells. In many countries (including the United States, European Union and Japan) Nivolumab is approved to treat certain cancer types. The purpose of the study is to test the safety and effectiveness of nivolumab in patients with advanced RCC when given intermittently.

Nivolumab is approved by the U.S. Food and Drug Administration (FDA) for the treatment of advanced kidney cancer, non small cell lung cancer, classical Hodgkin Lymphoma and Metastatic Melanoma. Nivolumab is FDA-approved for advanced RCC because has been shown to shrink RCC tumors that have spread outside the kidney.

DETAILED DESCRIPTION:
Primary Objective:

- To determine the feasibility of intermittent nivolumab therapy in patients with metastatic renal cell carcinoma.

Secondary Objectives:

* To determine the clinical outcome (overall response rate (ORR), progressive free survival (PFS), overall survival (OS)) in metastatic renal cell carcinoma patients treated with intermittent nivolumab therapy.
* To evaluate the toxicity of intermittent nivolumab therapy in patients with metastatic renal cell carcinoma.

Correlative Objective

- Investigate correlations between baseline and post-treatment immunomodulatory cells [specifically, myeloid-derived suppressor cells (MDSC) regulatory T cells (Treg), cluster of differentiation 4 (CD4) and cluster of differentiation 8 (CD8), T Cells, T-cell receptor (TCR) repertoire and time off therapy.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1:

  * Must have received at least one but not more than two prior anti-angiogenic therapy regimens (including, but not limited to, sunitinib, sorafenib, pazopanib, axitinib, tivozanib, and bevacizumab) in the advanced or metastatic RCC setting. Prior cytokine therapy (eg, IL-2, IFN-a), vaccine therapy, or treatment with cytotoxics is also allowed.
  * No more than three total prior systemic treatment regimens in the advanced or metastatic RCC setting.
* Cohort 2:

  --Achieved SD, PR, or CR after administration of front-line therapy with Ipi/Nivo (up to 4 doses) for advanced/metastatic RCC followed by 24 weeks (+/- 8 weeks; minimum 3 infusions) of Nivo maintenance. Patient enrollment will occur after completion of 24 weeks (+/- 8 weeks; minimum 3 infusions) of maintenance nivolumab.
* Histological confirmation of renal cell carcinoma (RCC) (any histology)
* Advanced or metastatic RCC.
* Measurable disease as defined by RECIST 1.1 criteria
* Must have received at least one but not more than two prior anti-angiogenic therapy regimens (including, but not limited to, sunitinib, sorafenib, pazopanib, axitinib, tivozanib, and bevacizumab) in the advanced or metastatic RCC setting. Prior cytokine therapy (for example, Interleukin (IL)-2, interferon (IFN)-α), vaccine therapy, or treatment with cytotoxics is also allowed.
* Patients treated with neoadjuvant and/or adjuvant therapy prior to development of metastatic disease may also be included provided that at least 12 months have elapsed since last dose. These regimens do not count toward total number of prior therapies permitted for trial inclusion.
* No more than three total prior systemic treatment regimens in the advanced or metastatic RCC setting, and must have evidence of progression on or after the last treatment regimen received and within 6 months prior to study enrollment.
* Karnofsky Performance Score (KPS) ≥70%
* Women of childbearing potential (WOCBP) must use effective method(s) of contraception have a negative serum or urine pregnancy test within 24 hours prior to the start of therapy, and must not be breastfeeding. Pregnant women are excluded from this study because animal studies have demonstrated that nivolumab can cause fetal harm when administered to pregnant women. Breastfeeding women are excluded from this study because nivolumab may be excreted in human milk and the potential for serious adverse reactions in nursing infants.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year
* Willing and able to provide informed consent.
* Laboratory criteria for study entry must meet the following criteria:

  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 40 mL/min (measured or calculated using the Cockcroft-Gault formula).
  * white blood cell count ≥ 2000/µL
  * Neutrophils ≥ 1500/µL
  * Platelets ≥ 100,000/µL
  * Hemaglobin ≥ 9.0g/dL
  * Aspartate Aminotransferase (AST) and alanine transaminase (ALT) ≤ 3.0 x ULN
  * Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)

Exclusion Criteria:

* Cohort 1 only:

  --Prior treatment with an anti-programmed death (PD)-1, anti-programmed death ligand 1 (PD-L1), anti-programmed death ligand 2 (PD-L2), anti-Cluster of differentiation (CD137), or anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Anti-cancer therapy less than 14 days prior to the first dose of study drug (less than 28 days for bevacizumab) or palliative, focal radiation therapy less than 14 days prior to the first dose of study drug.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Patients are excluded if they have active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if metastases have been treated and there is no imaging evidence of progression for 28 days after treatment is complete and within 28 days prior to the first dose of nivolumab administration.
* Major surgery (eg, nephrectomy) less than 28 days prior to the first dose of study drug.
* Any active known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition or prior therapy requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to the first dose of study drug. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
* Any known active chronic liver disease.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Any positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection.
* Known medical condition (for example, a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results.
* Strong Cytochrome P450 3A4 (CYP3A4) inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
the proportion of patients who receive intermittent therapy | Expected duration 5.5 months
  For cohort I: Assess feasibility of an intermittent dosing schedule, where feasibility is defined in terms of the proportion of patients eligible for intermittent therapy who actually receive it. An underlying acceptance rate of >80% is arbitrarily considered necessary in order to accept the intermittent schedule as feasible whereas an acceptance rate <50% is considered evidence that the intermittent schedule is not feasible
Rate of participants who maintain CR/PR off therapy for at least 9 months | Up to 9 months after treatment
  For cohort II: Rate of participants who maintain CR/PR off therapy for at least 9 months

SECONDARY OUTCOMES:
Change in tumor burden | Expected duration 5.5 months
Objective Response | Expected duration 5.5 months
  Number of patients with tumor response per the RECIST 1.1 Criteria:
  Complete response (CR) is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non target) must have reduction in short axis to <10 mm.
  Partial response (PR) is defined as a greater than or equal to 30% decrease in the sum of the longest dimensions of the target lesions
  Progressive disease (PD) is defined as a greater than or equal to 20% increase in the sum of the longest dimensions of the target lesions, or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Stable disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
Length of Progression Free Survival | Expected duration 5.5 months
  Time from enrollment in the study to progression, when progression is defined as a greater than or equal to 20% increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Percent of patients who experience grade 3 AE or higher with re-induction ipi/nivo | up to 100 days after end of treatment
  Estimate toxicity rate in participants undergoing reinduction with ipilimumab/nivolumab as measured by percent of patients who experience grade 3 AE or higher

CONTACTS AND LOCATIONS:
Overall Officials: Moshe C. Ornstein, MD, MA, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Ornstein MC, George L, Wei W, Diaz-Montero CM, Rayman P, Martin A, Basu A, Beckermann KE, Nizam A, Wee CE, Gilligan TD, Gupta S, Rini BI. Phase II Trial of Intermittent Therapy in Patients with Metastatic Renal Cell Carcinoma Treated with Front-line Ipilimumab and Nivolumab. Clin Genitourin Cancer. 2024 Dec;22(6):102181. doi: 10.1016/j.clgc.2024.102181. Epub 2024 Jul 31. PMID 39208489
- [Derived] Ornstein MC, Wood LS, Hobbs BP, Allman KD, Martin A, Bevan M, Gilligan TD, Garcia JA, Rini BI. A phase II trial of intermittent nivolumab in patients with metastatic renal cell carcinoma (mRCC) who have received prior anti-angiogenic therapy. J Immunother Cancer. 2019 May 16;7(1):127. doi: 10.1186/s40425-019-0615-z. PMID 31097024